CLINICAL TRIAL: NCT06781723
Title: Improving the Anabolic Action of Plant-based Foods Using Complementary Proteins
Acronym: CompProtein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0582; 7007302 (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2024-10-07; First posted 2025-01-17 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Health; Recreational Activities; Muscle Protein Synthetic Response to Protein; Muscle Protein Synthesis
Keywords: protein; metabolism; plant protein; vegan; protein synthesis; complementary proteins
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rice and Beans (COMP) (Experimental): Rice and Beans
  After resistance exercise, participants will ingest a meal of 123g Rice, 123g Black Beans (246 g; 575kcal, 20 g Protein, 121 g Carbohydrate, 0.7 g Fat, 1.78 g Fat)
  Interventions: Behavioral: Resistance Exercise; Other: Rice and Beans
- Isolated Nutrients (ISO) (Active Comparator): This condition is isonitrogenous and a similar nutrient profile to the experimental complementary mixed meal. The drink is comprised of crystalline amino acids, carbohydrate, fat, and fiber that is matched to rice and beans meal composition.
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: Isolated Mixture

INTERVENTIONS:
Behavioral: Resistance Exercise — Participants will perform leg press and leg extension immediately prior to ingestion of rice and beans or isolated mixture.
Dietary Supplement: Isolated Mixture — Participants will ingest isolated mixture of crystalized amino acids, maltodextrin, fiber and oil immediately after resistance exercise.
  Other Names: ISO
  Arms: Isolated Nutrients (ISO)
Other: Rice and Beans — Participants will ingest cooked rice and beans meal immediately after resistance exercise.
  Arms: Rice and Beans (COMP)

SUMMARY:
In a crossover design 10 young healthy adults (20-35 y) will receive stable isotope tracer infusions and perform a single bout of resistance exercise. Immediately after exercise participants will ingest either 246 g of rice and beans or its constituent macronutrients as isolated amino acids, carbohydrates, fiber, and fat. Repeated blood and muscle biopsies will be collected to determine amino acid concentrations, anabolic signaling and myofibrillar protein synthesis rates during the trials.

DETAILED DESCRIPTION:
1. Preliminary Testing Preparation: Participants will arrive for the preliminary testing session after an overnight fast (~10 h no caloric foods/beverages consumed) and having refrained from exercise for the 72 h prior. Prior to any in-person procedures, participants will be briefed on the procedures and risks associated with participation via reviewing the informed consent document. Participants will be encouraged to ask questions and have their questions answered prior to being asked if they'd like to continue. Confirmation will be documented via signature on an informed consent process form.

   1.1 Anthropometrics: Upon provision of consent, participants' height and weight will be measured to confirm body mass index (BMI) is within eligibility limits (18.5 - 30 kg/m^2). Since participants have already been assessed for all other inclusion and exclusion criteria, an eligible BMI will result in study inclusion and continuation of the preliminary testing session. Following confirmation of study eligibility, blood pressure will be measured by a trained member of the research team. Subsequently, body composition will be determined via dual energy x-ray absorptiometry (DEXA) in accordance with manufacturer recommendations. Briefly, participants will be asked to remove all metal objects from their person prior to being positioned by a trained technician for accurate measurement of lean body mass and fat mass. The scan lasts approximately 6-10 minutes during which the participant will be instructed to remain motionless.

   1.2 Resting Metabolic Rate: Resting metabolic rate (RMR) will be assessed via indirect calorimetry. This is a non-exertional test whereby RMR is measured using an automated gas analysis system. This device measures oxygen consumption and carbon dioxide production as the difference between inspired and expired gas concentrations. Prior to the beginning of the test, participants will lie supine on a table and a clear, hard plastic hood and soft, clear plastic drape will be placed over the participants neck, head, and shoulders to capture expired gases. Participants will then lie motionless without falling asleep while respiratory gas concentrations are captured. Testing will conclude when RMR is stable for at least 20 min (typically ~30 min from the onset).

   1.3 Ten-Repetition Maximum (10RM) Testing: Following resting metabolic rate testing, participants will have their 10RM tested for the leg extension and leg press. To begin, participants will cycle at a self-selected pace on a standard cycle ergometer for ~5 minutes. Participants will then complete a set of 8-10 repetitions at ~50% of their predicted 10RM followed by 1-2 minutes of rest. The load will then be set at ~90% of their predicted 10RM. Load will be increased by 2.5-5.0% following each successful attempt until failure (typically within 5 attempts). Two minutes of rest will be allotted between maximal attempts and 5 minutes between exercises. Leg extension will be tested first followed by leg press. Before leaving the laboratory, participants will be allowed to ask any questions they have before concluding the session.

   1.4 Habitual Diet Record: Current diet intake will be assessed through an online automated self-administered (ASA24) diet record system. Participants will receive their individual and private username and password. They will be asked to record 3 consecutive days (2 weekdays, 1 weekend day). As it is an online system, they can complete off-site, at their leisure.

   1.5 Planning: Prior to leaving the laboratory, participants and the research team will identify a date for the first infusion trial (at least 7 days following preliminary testing). Moreover, the research team will provide participants with a standardized meal to consume the night before the first infusion and instructions to refrain from strenuous exercise and alcohol consumption for 72 and 24 hours leading into the first trial. Participants will also be offered a snack prior to leaving the laboratory.
2. Infusion Trials

2.1 Preparation: At least 7 days following preliminary testing or the previous infusion, participants will be asked to return to the laboratory for an infusion trial. On the morning of each infusion, participants will arrive to the laboratory in the morning following an overnight (~10 h no caloric foods/beverages consumed) fast and having refrained from strenuous exercise and alcohol consumption for 72 and 24 hours, respectively. For 3 days preceding each trial, participants will be asked to record their dietary intakes via and online automated self-administered (24 hour) dietary record system (ASA24).

2.2 Stable Isotope Infusion: Upon arrival to the laboratory, participants will lay supine on a clinic-style bed before having an intravenous catheter placed into a dorsal hand or arm vein. No more than four attempts will be made to set the catheter. Following baseline blood sampling, a priming dose of L-[ring-13C6]phenylalanine (2 μmol/kg) will be administered prior to initiation of a constant infusion (0.05 μmol/kg/min) using a calibrated infusion pump. The stable isotope amino acid tracers applied in this experiment are not radioactive and are completely safe. These stable isotopes will enrich the amino acid pool in the body allowing us to identify the rate of incorporation of amino acids into the tissues. The preparation of the tracers for intravenous administration will occur in a sterile environment under a laminar flow hood dedicated to the preparation of tracers and in accordance with Good Manufacturing Practices guidelines.

2.3 Blood Collection: Following initiation of the infusion, a second intravenous catheter will be placed in the contralateral side in a hand or arm vein for repeat blood sampling. Blood samples will be collected will be collected 12 times during the first infusion and 10 times during the second infusion. At time points that coincide with biopsy times (-150, -30 and 300 min), ~16 mL will be collected (7 mL plasma, 7 mL serum, and ~2 mL waste). At all other time points (-210, -90, 0, 30, 60, 90, 120, 180, and 240 min) ~9 mL will be collected (7 mL plasma and ~2 mL waste). Thus, the total volume collected during the first infusion and second infusion will be ~129 mL and ~104 mL, respectively. Blood will be collected into evacuated tubes using Leur-Lok access device connected to a 4-way stopcock. Between draws, the catheter will be kept patent using a saline drip at a low rate (~60 cc/hr).

2.4 Muscle Collection: A total of five muscle biopsies will be collected (three as a part of 1st infusion and two during 2nd infusion). The biopsy procedure involves removal of a small piece of muscle tissue using a sterile hollow needle (Bergström needle) and will be performed by Dr. Nicholas Burd under the auspices of Dr. Jared Willard, MD. Participants will rest on a bed and the area for the biopsy will be shaved, if required. Subsequently, the area will be sterilized using 4% chlorhexidine gluconate before 5 mL of local anesthetic (2% Xylocaine with 1:100,000 epinephrine) is injected subcutaneously with special care to avoid infiltrating the muscle. Once the anesthetic is active (~10 min), Dr. Burd will make a small incision (~4-5 mm) in the skin in order to create an opening through which to put the biopsy needle for tissue collection. Dr. Burd will quickly cut of a small piece of muscle (~50- 100 mg; about the size of a standard pencil eraser) and remove the needle from the subject's leg. During the sample collection (~30 sec), the subjects may feel a sensation of deep pressure in their leg. A sterile disposable drape will be placed under the participant's thigh and sterile gloves will be used for all biopsy procedures.

After the biopsy is completed, a trained research team member will apply pressure with sterile gauze until the bleeding stops (at least 10 min). Subsequently, the incision site will be closed using butterfly stitches (Steri-strips) following by application of a bandage. An elastic pressure wrap will be applied on top of the bandage in order to minimize the chance of bruising. Participants will then be instructed to leave the butterfly stitches and the pressure wrap on the wound for 96 and 24 hrs, respectively.

The participant will be provided with a "biopsy care kit" (described in section 10.1/Biopsy care kit) in order to properly care for the incision after leaving the laboratory. A member of the research team will contact the participants in the day following the trial to check on the healing process.

2.5 Resistance Exercise and Meal Ingestion: Immediately following the closure of the second biopsy in the first infusion trial and after the closure of first biopsy in the second trial participants will begin warming up for an acute bout of resistance exercise. To begin, participants will cycle at a self-selected pace on a standard cycle ergometer for 5 minutes. Subsequently, participants will begin resistance exercise. Participants will complete a warmup set at ~60% of their ten-repetition maximum (10RM) measured at preliminary testing followed by 4 sets of 10-12 repetitions at ~90% 10RM with 1-3 minutes rest between sets for both leg extension and leg press. Participants will match the load, sets, and repetitions from the first infusion during their second trial.

Immediately following the completion exercise, participants will return to the infusion room to consume their meal. During their first infusion, participants will be randomly assigned to consume either 246 g of commercially available rice and black beans (~610 kcal; ~20 g protein, ~127 g of carbohydrate) or isocaloric and isonitrogenous drink of crystallized amino acids and maltodextrin. During their second trial, participants will be randomly assigned to consume the remaining condition.

Commercially-available rice and black beans will be separately cooked and mixed right before consumption on the infusion trial day. The meal will be cooked to an internal temperature of at least 160°F in accordance with the USDA's minimum internal temperature to prevent foodborne illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 yrs
* Pre-menopausal
* Recreationally-active
* Weight stable for prior 6 months

Exclusion Criteria:

Age outside of range (20 - 35 yrs)

* Pregnancy
* Irregular menstrual cycles (i.e., ~21 day or ~35 day cycle)
* Participation in previous research using [13C6]phenylalanine
* Participation in other ongoing research that interferes with this study (e.g., conflicting diet, activity interventions, etc.)
* Any hospitalization or surgery for a metabolic, cardiovascular, or neuromusculoskeletal complication within the past year
* Allergy or hypersensitivity to local anesthetics, latex, or adhesives (bandages, medical tape, etc.)
* Excess scarring after injury
* History of excess bleeding after cut
* Chronic or frequent dizziness/fainting, and arm or leg weakness/numbness
* Arthritis
* Tumors
* Mental Illness
* Hepatorenal, cardiovascular musculoskeletal, autoimmune, or neurological disease or disorder
* Predisposition to hypertrophic scarring or keloid formation
* Physical activity limitations
* Consumption of ergogenic-levels of dietary supplements that may affect muscle mass (e.g., creatine, HMB), insulin-like substances, or anabolic/catabolic pro-hormones (e.g., DHEA) within 6 weeks prior to participation
* Consumption of thyroid, androgenic, or other medications known to affect endocrine function
* Consumption of medications known to affect protein metabolism (e.g., prescription-strength corticosteroids, non-steroidal anti-inflammatories, or acne medication)
* Unwillingness to comply with study procedures
* Weight unstable (variation >5% of bodyweight in last 6-12 months)
* Current or previous tobacco use with last 6 months
* Obesity (body mass index; BMI >>30 kg∙m^-2)
* Score of less than 14 on the Godin-Shephard Leisure-Time Physical Activity Questionnaire
* Phenylketonuria
* Anyone hospitalized previously for COVID-19 without a cardiovascular workup screening for cardiovascular issues post-infection
* Anyone recovering from COVID-19 infection within the preceding 10 days

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein fractional synthesis rate | Basal FSR (from -150 to - 30 min), Postprandial FSR (from -30 to 300min)
  Myofibrillar protein synthesis rates will be assessed during the postabsorptive and postprandial periods of experimental primed-constant stable isotope infusions.
Plasma Amino Acid Concentrations | Post absorptive (-210, -150, -90, -30, 0 min); Post prandial (30, 60, 90, 120, 180, 240, 300 min)
  Amino acid concentrations will be assessed in the postabsorptive state (-210, -150, -90, -30, 0 min) and postprandial state (30, 60, 90, 120, 180, 240, 300 min) via LC/MS/MS.

SECONDARY OUTCOMES:
Activation of Anabolic Signaling Targets | -150 min, -30 min, 300 min
  Phosphorylation of mTOR-dependent anabolic signaling targets will be assessed via Western Blotting (phosphorylated-to-total ratio).

CONTACTS AND LOCATIONS:
Locations (1):
- Louise Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Because it is not planned to published in any ICMJE journal.